CLINICAL TRIAL: NCT03586752
Title: "iGOGO-Automated External Defibrillator Donation "Continuing Education Project
Brief Title: CPR Education: Traditional Program Versus On-line Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GMRPG3F1273
Record Dates: First submitted 2018-06-28; First posted 2018-07-16 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: HQCPR between standard and on-line program; Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On-line group (Experimental): On-line program course
  Interventions: Other: On-line program
- Standard group (Active Comparator): Standard program course
  Interventions: Other: Standard program

INTERVENTIONS:
Other: On-line program — 18 minutes on-line video at home and 30 minutes CPR skill practice at scene in 3 days after watching on-line video
  Arms: On-line group
Other: Standard program — 60-minute CPR teaching video with practice, 20 minutes of automated electrical defibrillator operation, and a 10-minute discussion with regard to the legal issues associated with bystander CPR in Taiwan
  Arms: Standard group

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) is an important public health issue. Chang Gung Memorial Hospital, a university affiliated medical center in Taoyuan city, northern Taiwan, actively cooperated with the government policy to donate a total of 250 automated external defibrillators (AED) and to deploy them in public areas during the period of 2012 to 2014. In addition, nearly 200 courses of cardiopulmonary resuscitation (CPR) education for healthcare providers and citizens were provided.

In order to keep the skills and the abilities of emergency medical responses in these 200 and more AED recipient areas, repeated CPR education and training should be implemented. Quality assurance and regular follow-up by medical directors with professional advice and feedback can therefore be provided at the same time. Therefore, this project aims to assess the quality of emergency responses in the recipient units in the next four years via regular follow-up by medical directors with advice and feedback. Continuing medical education of both e-learning and classes, online registration system, as well as first aid supplies will be provided at the regular follow-up visits. The results of this project will provide a feasible model of quality assurance of first aid and AED implementation program in the community.

DETAILED DESCRIPTION:
The core value of the investigation is to provide high quality, convenient, time-saving, and cost-effective CPR training model. The training proctors will either instruct laypersons or healthcare providers to watch on-line video for 18 minutes at home then practice the skills for 30 minutes in the training scene or provide standard CPR program (90 minutes in the scene) and empower them with the life-saving skills of CPR. The American Heart Association's CPR with a DVD and laerdal QCPR manikin will be used to record. Participants will be randomly allocate into either the on-line or standard method of the training program. To assess the effects of training, the participants will receive written examinations before and after the course. The investigators will also follow up with the study participants and conduct CPR skills tests at 6 and 12 months from the time of training to assess whether the subjects retain their skills or if they have an opportunity to use the skills that they learned. Information about the willing of performing CPR and satisfaction to the training will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 and over
* Adults who have not attended CPR training for at least one year prior to enrollment

Exclusion Criteria:

* unable to kneel to practice CPR
* pregnant
* unwilling to sign informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 832 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Written test for knowledge about CPR | 4 days
  Knowledge about CPR will be assessed via a written test before and after the CPR training. The test includes 25 questions with a total score of 100 (4 points for each).
CPR flow checklist | 4 days
  An evaluator who is blinded to the training allocation will assess the performance of CPR via a flow checklist. A total of 20 items will be checked with a maximum sum score of 40 points.

SECONDARY OUTCOMES:
The percentage of correct depth of all compressions | 90 minutes
  The percentage of correct depth (5-6 centimeters) of all compressions will be assessed by High Quality CPR (HQCPR).
  HQCPR is a machine with interactive response system which can provide information while performing CPR on manikin (Laerdal, Resusci Anne QCPR).
The percentage of correct speed of compressions of all compressions | 90 minutes
  The percentage of correct speed of compressions (100 to 200 per minute) of all compressions will be assessed by HQCPR.
  HQCPR is a machine with interactive response system which can provide information while performing CPR on manikin (Laerdal, Resusci Anne QCPR).
The percentage of correct recoil of all compressions | 90 minutes
  The percentage of correct recoil (full chest recoil) of all compressions will be assessed by HQCPR.
  HQCPR is a machine with interactive response system which can provide information while performing CPR on manikin (Laerdal, Resusci Anne QCPR).
The average compression depth | 90 minutes
  The average compression depth (unit in centimeter) is calculated by summing up the depth of each compression then to be divided by the number of total compressions. The compression depth is recorded by HQCPR.
  HQCPR is an interactive response machine to provide the information on depth, speed and recoil while performing CPR on manikin (Laerdal, Resusci Anne QCPR).
The average compression speed | 90 minutes
  The average compression speed is presented as the number of compressions per minute by HQCPR.
  HQCPR is an interactive response machine to provide the information on depth, speed and recoil while performing CPR on manikin (Laerdal, Resusci Anne QCPR).

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Yu Chien, Dr., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chien CY, Fang SY, Tsai LH, Tsai SL, Chen CB, Seak CJ, Weng YM, Lin CC, Chien WC, Huang CH, Lin CY, Chaou CH, Liu PH, Tseng HJ, Chen JC, Peng SY, Cheng TH, Hsu KH, Ng CJ. Traditional versus blended CPR training program: A randomized controlled non-inferiority study. Sci Rep. 2020 Jun 22;10(1):10032. doi: 10.1038/s41598-020-67193-1. PMID 32572100